CLINICAL TRIAL: NCT04688255
Title: Randomized Controlled Trial Using Telehealth-delivered Rehabilitative Exercise to Treat Youth With Prolonged Concussion Recovery (Mobile Subthreshold Exercise Program, MSTEP-R01)
Brief Title: Mobile Subthreshold Exercise Program for Concussion--R01
Acronym: MSTEP-R01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Sara PD Chrisman, MD MPH, Associate Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00002697; 1R01HD094722-01A1 (NIH)
Record Dates: First submitted 2020-12-23; First posted 2020-12-29 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Concussion, Brain; Concussion, Mild; Brain Injuries, Traumatic; Persistent Post Traumatic Headache; Post-Concussion Syndrome; Post-Concussive Syndrome, Chronic
Keywords: Traumatic brain injury; Concussion; Exercise; Physical activity; Subthreshold; Treatment; Pediatric; Child
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Post-Concussion Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT)
Who Masked: Participant, Outcomes Assessor
Masking Description: Using an active control (stretching) and both arms described as exercise intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (MSTEP) (Experimental): REHABILITATIVE EXERCISE: Participants will be asked to exercise at home daily for 6 weeks, meeting with an RA weekly via video conference to gradually increase the intensity and duration of exercise based on symptom tolerance. The eventual goal will be to achieve 60 minutes of MVPA daily (US Federal recommendations). They will wear a personal fitness device (Fitbit) to track whether they are achieving their HR goals.
  Interventions: Behavioral: MSTEP
- Control group (Stretching) (Active Comparator): STRETCHING: Participants will be asked to complete stretches daily. They will initially be given two stretches, primarily focused on the neck and upper back. Additional stretches will be added through weekly discussions with the study RA.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: MSTEP — Aerobic exercise that is advanced weekly
  Arms: Intervention group (MSTEP)
Behavioral: Stretching — Stretching exercises that are advanced weekly
  Arms: Control group (Stretching)

SUMMARY:
Approximately 1.9 million youth sustain a concussion each year, and up to 30% experience persistent post-concussive symptoms (PPCS) such as headache, dizziness, and difficulty focusing that continue for weeks or months. PPCS results in greater utilization of sub-specialty care and can impact immediate and long-term social development, cognitive function and academic success. Previous recommendations for treating PPCS have focused on cognitive and physical rest, but more recently guidelines have shifted based on new research suggesting the benefit of rehabilitative exercise for PPCS. The rationale behind using exercise to treat youth with concussion is that gradually increasing physical activity facilitates return to full function. Rehabilitative exercise has since become one of the most common approaches to treating youth with PPCS, but access is challenging since most programs require weekly centralized visits with a concussion specialist. To bridge this gap, the investigators developed a telehealth-delivered approach to treat PPCS, utilizing physical activity trackers (Fitbits) and weekly video conferences with trained research staff. They then conducted a series of pilot studies with this approach, finding excellent feasibility, acceptability, and evidence for more rapid declines in concussive symptoms compared to controls. The investigators also found preliminary evidence that mechanisms behind this intervention may stem from both physiologic processes due to increased moderate-to-vigorous physical activity (MVPA) and psychologic processes such as reducing fear- avoidance of concussive symptoms. They now propose a fully-powered randomized controlled trial (RCT) to asses the efficacy of the "Mobile Subthreshold Exercise Program" (M-STEP) for treating youth with PPCS.

DETAILED DESCRIPTION:
The investigators will recruit n=200 youth 11-18 years old with PPCS. Youth will be randomized to 6 weeks of either usual care plus M-STEP (intervention) or usual care plus stretching (control). Youth in M-STEP will be coached through gradual increases in intensity and duration of rehabilitative exercise via weekly video conferencing (Zoom) and will use Fitbits to guide their progress. Youth in the stretching group will act as attention controls. All youth will complete research-grade measures at multiple time points. Youth will be followed for a total of 6 months. Data will be analyzed using mixed effects models to examine differences between experimental groups in the primary outcome, trajectory of concussive symptoms, and the secondary outcome, changes over time in health-related quality of life, on an intention-to-treat basis. Potential mediators of the treatment effect will also be examined, including fear-avoidance of concussive symptoms and MVPA, and explore the impact of factors such as patient sex and parental protective behaviors.

The investigators thus assert the following hypotheses:

Hypothesis 1: M-STEP youth will have more rapid declines in HBI and improvement in PedsQL compared to control youth

Hypothesis 2: M-STEP youth will have greater increases in MVPA over time than control youth, and these increases will predict more rapid improvement in HBI and PedsQL.

Hypothesis 3: M-STEP youth will have steeper declines in fear-avoidance compared to control youth, and these declines will predict more rapid improvement in HBI and PedsQL.

IMPACT: The proposed study will definitively answer the question of whether a mobile sub-threshold exercise program (M-STEP) improves outcomes for youth with PPCS. It will also provide essential information about both the long-term impact of this intervention and potential mediators as well as biopsychosocial factors that influence treatment response. The study design uses a rigorous protocolized smartphone administered mHealth intervention that will be readily reproducible and generalizable to the majority of youth with PPCS. If successful, this will be one of the few evidenced-based interventions available to treat youth with PPCS.

ELIGIBILITY:
Inclusion Criteria:

* Youth 11-18 years
* Concussion occurring 1 week to 12 months prior to the start of the study and diagnosed by a clinician trained in concussion management consistent with the 2017 Berlin consensus definition of concussion ("A traumatic brain injury, induced by biomechanical forces")
* Persistent post-concussive symptoms as defined by the presence of at least 3 concussive symptoms rated at least 2 or greater on the Health and Behavior Inventory (HBI) and a total score of at least 10
* Can be located anywhere as all study procedures are remote

Exclusion Criteria:

* Youth not fluent in English or at least one Parent not fluent in English or Spanish
* Other injuries or medical conditions in addition to concussion that have prompted a clinician to recommend against MVPA, such as concerning abnormalities on routine brain imaging
* Youth who indicate that they are completing an average of 30 minutes per day or greater of physical activity that increases their heart rate (indicative of a minimal need for a physical activity intervention)
* Youth who have previously engaged with a Physical Therapist to increase aerobic activity
* Youth who have been fully cleared for sport

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Concussive symptoms (Health Behavior Inventory, HBI)--youth, a 21 item 0-3 likert scale with higher scores indicating more severe symptoms | Baseline, weekly during the intervention (x6 weeks), 3 months and 6 months.
  Examine trajectory of concussive symptoms over time. The central hypothesis is that the intervention group will have a more rapid decline in concussive symptoms..
Pediatric Quality of Life (PEDsQL, parent and youth), a 23 item 0-4 likert scale that is scaled to 0-100 with higher scores indicating better function | Baseline, 6 weeks, 3 months and 6 months.
  Examine trajectory of concussive symptoms over time. The central hypothesis is that the intervention group will have a more rapid improvement in health-related quality of life.

SECONDARY OUTCOMES:
Fear of Pain Questionnaire (FOPQ, parent and youth), adapted for concussive symptoms, 24 item (child) and 23 item (parent) 0-4 likert scales with higher scores indicating greater fear-avoidance | Baseline, 6 weeks, 3 months and 6 months.
  Examine trajectory of fear-avoidance over time and assess for mediation of change in concussive symptoms. The central hypothesis is that decreases in fear-avoidance of concussive symptoms will partially mediate the decline in concussive symptoms.
Moderate-Vigorous Physical Activity (MVPA), measured with hip-mounted actigraphy | Baseline, 6 weeks, 3 months
  Examine trajectory of MVPA over time and assess for mediation of change in concussive symptoms. The central hypothesis is that increases in MVPA will partially mediate the decline in concussive symptoms.

OTHER OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9), standardized measure of depressive symptoms, a 9-item 0-3 likert scale with higher scores indicating more severe symptoms | Baseline, 6 weeks, 3 months, 6 months
  Explore trajectory of depressive symptoms during the intervention. The central hypothesis is that depressive symptoms will decline during the intervention.
Generalized Anxiety Disorder Scale-7 (GAD-7), standardized measure of anxiety symptoms, a 7-item 0-3 likert scale with higher scores indicating more severe symptoms | Baseline, 6 weeks, 3 months, 6 months
  Explore trajectory of anxiety symptoms during the intervention. The central hypothesis is that anxiety symptoms will decline during the intervention.
Adolescent Sleep Wake Scale (ASWS)-10, standardized survey (self-report) regarding sleep quality, a 10-item 0-5 likert scale reported as the mean with higher scores indicating improved sleep quality | Baseline, 6 weeks, 3 months, 6 months
  Explore trajectory of self-reported sleep quality during the intervention. The central hypothesis is that sleep quality will improve during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sara P Chrisman, MD MPH, Principal Investigator — University of Washington and Seattle Children's Hospital
Locations (1):
- Seattle Childrens Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chrisman SPD, Whitlock KB, Mendoza JA, Burton MS, Somers E, Hsu A, Fay L, Palermo TM, Rivara FP. Pilot Randomized Controlled Trial of an Exercise Program Requiring Minimal In-person Visits for Youth With Persistent Sport-Related Concussion. Front Neurol. 2019 Jun 17;10:623. doi: 10.3389/fneur.2019.00623. eCollection 2019. Erratum In: Front Neurol. 2020 Feb 21;11:6. doi: 10.3389/fneur.2020.00006. PMID 31316446
- [Background] Chrisman SPD, Whitlock KB, Somers E, Burton MS, Herring SA, Rowhani-Rahbar A, Rivara FP. Pilot study of the Sub-Symptom Threshold Exercise Program (SSTEP) for persistent concussion symptoms in youth. NeuroRehabilitation. 2017;40(4):493-499. doi: 10.3233/NRE-161436. PMID 28222566
- [Derived] Chrisman SPD, Zhou C, Sahlberg J, Bollinger BJ, Hansen C, Mendoza JA, Brooks MA, Rivara FP, Palermo TM. Psychometrics of a fear-avoidance measure adapted for youth with persistent postconcussive symptoms: Fear of Concussive Symptoms Questionnaire (FOCSQ) child and parent-proxy versions. Neuropsychology. 2025 Oct 2. doi: 10.1037/neu0001031. Online ahead of print. PMID 41037445
- [Derived] Chrisman SPD, Bollinger BJ, Mendoza JA, Palermo TM, Zhou C, Brooks MA, Rivara FP. Mobile Subthreshold Exercise Program (MSTEP) for concussion: study protocol for a randomized controlled trial. Trials. 2022 Apr 26;23(1):355. doi: 10.1186/s13063-022-06239-3. PMID 35473570